CLINICAL TRIAL: NCT02667483
Title: Phase I/II Study of DS-5141b: Open-label Study of DS-5141b in Patients With Duchenne Muscular Dystrophy
Brief Title: Study of DS-5141b in Patients With Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS5141-A-J101; 153072 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-07

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; DMD; Oligonucleotides, Antisense; Exon skipping
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DS-5141b (Experimental): DS-5141b, Subcutaneous injection
  Part 1: DS-5141b will be injected subcutaneously once a week for 2 weeks at the following dose levels. Dose escalation will be performed. DS-5141b will be administered at dose levels 1 and 3 in Cohort 1 and at dose levels 2 and 4 in Cohort 2.
  * Level 1: 0.1 mg/kg
  * Level 2: 0.5 mg/kg
  * Level 3: 2.0 mg/kg
  * Level 4: 6.0 mg/kg
  Part 2: Two doses of DS-5141b will be selected based on the results obtained in Part 1. Each selected dose will be administered subcutaneously once a week for 12 weeks.
  Part 2-Extension-2: Two doses, 2.0 mg/kg or 6.0 mg/kg, of DS-5141b will be administered subcutaneously once a week for 48 weeks.
  Interventions: Drug: DS-5141b

INTERVENTIONS:
Drug: DS-5141b — DS-5141b, Subcutaneous injection

SUMMARY:
This is a phase I/II study to evaluate the safety, tolerability, efficacy, and pharmacokinetic (PK) profile of DS-5141b in patients with Duchenne muscular dystrophy (DMD) amenable to exon 45 skipping and to determine the dosage for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of out-of-frame deletion(s) that could be corrected by dystrophin gene exon 45 skipping.
* Intact muscles of adequate quality for biopsy to allow evaluation of the efficacy of the study drug.
* Boys aged from 5 years to <11 years.
* Patients able to walk at least 325 meters in the 6-minutes walk test.
* Glucocorticoid-naive patients, or patients who have used glucocorticoids for at least 6 months prior to enrollment in this study with no dose changes for at least 3 months prior to enrollment.

Exclusion Criteria:

* A genetic mutation that can not be expected the expression of dystrophin protein by dystrophin gene exon 45 skipping.
* A concurrent illness other than DMD that can cause muscle weakness and/or impairment of motor function.
* Current or history of severe disorder.
* Left ventricular ejection fraction (LEVF) <55%.
* Corrected QT interval (QTc) >0.45 sec.

Ages: 5 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (2):
- Japan (2):
  - Kobe University Hospital, Hyōgo, Kobe-shi
  - National Center of Neurology and Psychiatry, Tokyo, Kodaira-shi

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants were screened; 8 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 2 clinic centers in Japan.
Groups:
- DS-5141b 2.0 mg/kg: All participants who received a subcutaneous injection of DS-5141b 2.0 mg/kg once a week.
- DS-5141b 6.0 mg/kg: All participants who received a subcutaneous injection of DS-5141b 6.0 mg/kg once a week.
Period: Overall Study
Arm/Group | DS-5141b 2.0 mg/kg | DS-5141b 6.0 mg/kg
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | DS-5141b 2.0 mg/kg | DS-5141b 6.0 mg/kg | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 5 | 8
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.3 (1.5) | 7.2 (1.9) | 6.9 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting at Least One Treatment-emergent Adverse Event (TEAE) In Participants With Duchenne Muscular Dystrophy
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event that emerges during treatment having been absent prior to treatment or reemerges during treatment or worsens in severity during treatment.
Time Frame: 48 Weeks of Part 2-Extension-2
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- All: DS-5141b 2.0 mg/kg: Participants who received a subcutaneous injection of DS-5141b 2.0 mg/kg once a week.
- All: DS-5141b 6.0 mg/kg: Participants who received a subcutaneous injection of DS-5141b 6.0 mg/kg once a week.
Arm/Group | All: DS-5141b 2.0 mg/kg | All: DS-5141b 6.0 mg/kg
Number analyzed (Participants) | 3 | 5
Participants | 3 | 5

2. Primary Outcome: Pharmacokinetic Parameter Maximum Concentration (Cmax) of DS-5141a (Free Form of DS-5141b) in Participants With Duchenne Muscular Dystrophy
Description: Pharmacokinetic parameters were assessed using non-compartmental methods.
Time Frame: Week 48 of Part 2-Extension-2
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | All: DS-5141b 2.0 mg/kg | All: DS-5141b 6.0 mg/kg
Number analyzed (Participants) | 3 | 5
ng/mL | 1320 (293) | 5190 (2590)

3. Primary Outcome: Pharmacokinetic Parameter Area Under the Curve (AUC) Tau of DS-5141a (Free Form of DS-5141b) in Participants With Duchenne Muscular Dystrophy
Description: Pharmacokinetic parameters were assessed using non-compartmental methods.
Time Frame: Week 48 of Part 2-Extension-2
Population: Pharmacokinetic parameters were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | All: DS-5141b 2.0 mg/kg | All: DS-5141b 6.0 mg/kg
Number analyzed (Participants) | 3 | 4
ng*h/mL | 23100 (5920) | 102000 (45600)

4. Primary Outcome: Pharmacokinetic Parameter Time to Maximum Concentration (Tmax) of DS-5141a (Free Form of DS-5141b) in Participants With Duchenne Muscular Dystrophy
Description: Pharmacokinetic parameters were assessed using non-compartmental methods.
Time Frame: Week 48 of Part 2-Extension-2
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | All: DS-5141b 2.0 mg/kg | All: DS-5141b 6.0 mg/kg
Number analyzed (Participants) | 3 | 5
hours | 1.98 [1.88 to 4.10] | 4.07 [3.93 to 8.00]

5. Primary Outcome: Pharmacokinetic Parameter Half-life (T1/2) of DS-5141a (Free Form of DS-5141b) in Participants With Duchenne Dystrophy
Description: Pharmacokinetic parameters were assessed using non-compartmental methods.
Time Frame: Week 48 of Part 2-Extension-2
Population: Pharmacokinetic parameters were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | All: DS-5141b 2.0 mg/kg | All: DS-5141b 6.0 mg/kg
Number analyzed (Participants) | 0 | 1
hours |  | 32.4

6. Primary Outcome: Mean Dystrophin Protein Expression in Muscle Tissue
Time Frame: Week 48 of Part 2-Extension-2
Population: Dystrophin protein expression was assessed in the Efficacy Analysis Set.
Measure: Mean (Standard Deviation); unit: percent of normal protein expression
Arm/Group | All: DS-5141b 2.0 mg/kg | All: DS-5141b 6.0 mg/kg
Number analyzed (Participants) | 3 | 5
percent of normal protein expression
  Baseline: Normalized by myosin heavy chain | 2.51 (4.13) | 1.86 (1.95)
  Post Extension Treatment: Normalized by myosin heavy chain | 3.65 (5.98) | 2.43 (2.42)

7. Secondary Outcome: Number of Participants With Exon 45-skipped Dystrophin mRNA Expression in Muscle Tissue Posttreatment
Time Frame: Week 48 of Part 2-Extension-2
Population: Dystrophin mRNA expression was assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | All: DS-5141b 2.0 mg/kg | All: DS-5141b 6.0 mg/kg
Number analyzed (Participants) | 3 | 5
Participants | 3 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline up to 48 weeks post extension period.
Arm/Group | DS-5141b 2.0 mg/kg | DS-5141b 6.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/5
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-5141b 2.0 mg/kg (N=3) | DS-5141b 6.0 mg/kg (N=5)
Appendicitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-5141b 2.0 mg/kg (N=3) | DS-5141b 6.0 mg/kg (N=5)
Appendicitis (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 2
Molluscum contagiosum (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 3
Otitis media (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Enuresis (Psychiatric disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Chalazion (Eye disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 2 | 0
Hypermetropia (Eye disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Growing pains (Musculoskeletal and connective tissue disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 1
Spontaneous penile erection (Reproductive system and breast disorders) | 0 | 1
Injection site bruising (General disorders) | 1 | 0
Injection site reaction (General disorders) | 3 | 5
Pyrexia (General disorders) | 2 | 1
Injection site discolouration (General disorders) | 1 | 2
Activated partial thrombroplastin time prolonged (Investigations) | 0 | 1
Albumin urine present (Investigations) | 1 | 2
Beta 2 microglobulin urine increased (Investigations) | 2 | 3
Beta-N-acetyl-D-glucosaminidase increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 0 | 1
Blood iron decreased (Investigations) | 0 | 2
Blood pressure diastolic increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0
Glucose urine (Investigations) | 0 | 1
Glucose urine present (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Monocyte count decreased (Investigations) | 0 | 1
Serum ferritin decreased (Investigations) | 0 | 2
Urinary casts (Investigations) | 1 | 1
White blood cell count increased (Investigations) | 1 | 1
Urinary sediment present (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 2
Urine albumin/creatinine ratio increased (Investigations) | 1 | 0
Urine ketone body present (Investigations) | 1 | 0
Cystatin C increased (Investigations) | 1 | 2
Alpha 1 microglobulin increased (Investigations) | 0 | 5
Magnetic resonance imaging brain abnormal (Investigations) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT02667483/Prot_SAP_000.pdf